CLINICAL TRIAL: NCT01824693
Title: A Randomized Phase II Study Comparing Two Different Conditioning Regimens Prior to Allogeneic Hematopoietic Cell Transplantation (HCT) for Children With Juvenile Myelomonocytic Leukemia (JMML)
Brief Title: Busulfan, Cyclophosphamide, and Melphalan or Busulfan and Fludarabine Phosphate Before Donor Hematopoietic Cell Transplant in Treating Younger Patients With Juvenile Myelomonocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASCT1221; NCI-2013-00738 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ASCT1221; ASCT1221; ASCT1221 (Other: Childrens Oncology Group); ASCT1221 (Other: CTEP); U10CA180886 (NIH); U10CA098543 (NIH)
Record Dates: First submitted 2013-04-02; First posted 2013-04-05 (Estimated); Results first posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Juvenile Myelomonocytic Leukemia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Juvenile | interventions — Busulfan; Cyclophosphamide; fludarabine phosphate; Melphalan; Mycophenolic Acid; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (busulfan, cyclophosphamide, melphalan) (Experimental): CONDITIONING REGIMEN: Patients receive busulfan IV QD, every 12 hours, or every 6 hours over 2-3 hours on days -8 to -5, cyclophosphamide IV QD over 60 minutes on days -4 and -3, and melphalan IV over 15-30 minutes on day -1.
  TRANSPLANT: Patients undergo allogeneic HCT no sooner than 24 hours after the last dose of chemotherapy.
  Patients receive tacrolimus IV or PO on days -1 to 98 (related donor) or 180 (unrelated donor) and mycophenolate mofetil IV over 2 hours or PO every 8 hours on days 1-30 (related donor) or 45 (unrelated donor).
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Busulfan; Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis; Drug: Melphalan; Drug: Mycophenolate Mofetil; Other: Pharmacological Study; Drug: Tacrolimus
- Arm II (busulfan, fludarabine phosphate) (Experimental): CONDITIONING REGIMEN: Patients receive busulfan as in Arm I and fludarabine phosphate IV over 1 hour on days -5 to -2.
  TRANSPLANT: Patients undergo allogeneic HCT as in Arm I.
  Patients receive tacrolimus IV or PO on days -1 to 98 (related donor) or 180 (unrelated donor) and mycophenolate mofetil IV over 2 hours or PO every 8 hours on days 1-30 (related donor) or 45 (unrelated donor).
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Busulfan; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Other: Pharmacological Study; Drug: Tacrolimus

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic HCT
  Other Names: Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT
Drug: Busulfan — Given IV
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
  Arms: Arm I (busulfan, cyclophosphamide, melphalan)
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
  Arms: Arm II (busulfan, fludarabine phosphate)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine nitrogen mustard; Sarcoclorin; Sarkolysin; WR-19813
  Arms: Arm I (busulfan, cyclophosphamide, melphalan)
Drug: Mycophenolate Mofetil — Given IV or PO
  Other Names: Cellcept; MMF
Other: Pharmacological Study — Correlative studies
Drug: Tacrolimus — Given IV or PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic

SUMMARY:
This randomized phase II trial studies how well giving busulfan, cyclophosphamide, and melphalan or busulfan and fludarabine phosphate before donor hematopoietic cell transplant works in treating younger patients with juvenile myelomonocytic leukemia. Giving chemotherapy before a donor hematopoietic transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient, they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. It is not yet known whether giving busulfan, cyclophosphamide, and melphalan or busulfan and fludarabine phosphate before a donor stem cell transplant is more effective in treating juvenile myelomonocytic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare ? in a randomized fashion ? the day 100 treatment related mortality (TRM) incidence for two myeloablative conditioning regimens, busulfan-fludarabine (fludarabine phosphate) (BU-FLU) and busulfan-cyclophosphamide-melphalan (BU-CY-MEL), prior to hematopoietic cell transplant (HCT) for children with juvenile myelomonocytic leukemia (JMML), in order to determine the preferred regimen for future trials.

II. To compare ? in a randomized fashion ? the 18-month event-free survival (EFS) following two different myeloablative conditioning regimens (BU-FLU vs. BU-CY-MEL) prior to HCT for children with JMML, in order to determine the preferred regimen for future trials.

SECONDARY OBJECTIVES:

I. To determine the 18-month relapse incidence (RI) following two different myeloablative conditioning regimens (BU-FLU vs. BU-CY-MEL) prior to HCT for children with JMML.

II. To determine the graft failure rates following two different myeloablative conditioning regimens (BU-FLU vs. BU-CY-MEL) prior to HCT for children with JMML.

TERTIARY OBJECTIVES:

I. To determine the rates of severe toxicities (grade 3/4) at day 100 post-HCT between the two myeloablative conditioning regimens (BU-FLU vs. BU-CY-MEL).

II. To determine the rates of acute and chronic (at 18 months post-HCT) graft-versus-host disease (GVHD) following HCT using two different conditioning regimens (BU-FLU vs. BU-CY-MEL) in children with JMML.

III. To create a JMML-specific pre-HCT index to allow better risk-stratification of future patients.

IV. To determine the feasibility of assessing post-transplant disease burden by donor chimerism measurements and allele-specific polymerase chain reaction (PCR) in mononuclear and sorted cell subsets.

V. To validate gene expression and methylation classifiers predictive of relapse in patients with JMML.

VI. To comprehensively assess genetic and biochemical alterations amongst patients with JMML who are treated on this transplant protocol.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I:

CONDITIONING REGIMEN: Patients receive busulfan intravenously (IV) over 2-3 hours once daily (QD), every 12 hours, or every 6 hours on days -8 to -5, cyclophosphamide IV over 60 minutes QD on days -4 and -3, and melphalan IV over 15-30 minutes on day -1.

TRANSPLANT: Patients undergo allogeneic HCT on day 0.

Patients receive tacrolimus IV or orally (PO) on days -1 to 98 (related donor) or 180 (unrelated donor) and mycophenolate mofetil IV over 2 hours or PO every 8 hours on days 1-30 (related donor) or 45 (unrelated donor).

ARM II:

CONDITIONING REGIMEN: Patients receive busulfan as in Arm I and fludarabine phosphate IV over 30-60 minutes on days -5 to -2.

TRANSPLANT: Patients undergo allogeneic HCT as in Arm I.

Patients receive tacrolimus IV or PO on days -1 to 98 (related donor) or 180 (unrelated donor) and mycophenolate mofetil IV over 2 hours or PO every 8 hours on days 1-30 (related donor) or 45 (unrelated donor).

After completion of study treatment, patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a strong clinical suspicion of JMML, based on a modified category 1 of the revised diagnostic criteria; specifically, eligible patients must have all of the following:

  * Splenomegaly
  * Absolute monocyte count (AMC) > 1000/uL
  * Blasts in peripheral blood (PB)/bone marrow (BM) < 20%
* For the 7-10% of patients without splenomegaly, the diagnostic entry criteria must include all other features described above and at least 2 of the following criteria:

  * Circulating myeloid precursors
  * White blood cell (WBC) > 10,000/uL
  * Increased fetal hemoglobin (HgbF) for age
  * Sargramostim (GM-CSF) hypersensitivity OR, patients must have been previously diagnosed with JMML
* Patients must be previously untreated with HCT
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients with a known germline mutation of PTPN11 (Noonan?s Syndrome) are not eligible
* Patients with a known history of NF1 (Neurofibromatosis Type 1) and either

  * A history of a tumor of the central nervous system (astrocytoma or optic glioma), or
  * A malignant peripheral nerve sheath tumor with a complete remission of < 1 year are not eligible
* Human immunodeficiency virus (HIV) positive patients are not eligible

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2013-06-24 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Dvorak, Principal Investigator — Children's Oncology Group
Locations (50):
- United States (44):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Norton Children's Hospital, Louisville, Kentucky
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (4):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
- Starship Children's Hospital, Grafton, Auckland, New Zealand

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Busulfan, Cyclophosphamide, Melphalan): CONDITIONING REGIMEN: Patients receive busulfan IV QD, every 12 hours, or every 6 hours over 2-3 hours on days -8 to -5, cyclophosphamide IV QD over 60 minutes on days -4 and -3, and melphalan IV over 15-30 minutes on day -1.
  TRANSPLANT: Patients undergo allogeneic HCT no sooner than 24 hours after the last dose of chemotherapy.
  Patients receive tacrolimus IV or PO on days -1 to 98 (related donor) or 180 (unrelated donor) and mycophenolate mofetil IV over 2 hours or PO every 8 hours on days 1-30 (related donor) or 45 (unrelated donor).
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo allogeneic HCT
  Busulfan: Given IV
  Cyclophosphamide: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Melphalan: Given IV
  Mycophenolate Mofetil: Given IV or PO
  Pharmacological Study: Correlative studies
  Tacrolimus: Given IV or PO
- Arm II (Busulfan, Fludarabine Phosphate): CONDITIONING REGIMEN: Patients receive busulfan as in Arm I and fludarabine phosphate IV over 1 hour on days -5 to -2.
  TRANSPLANT: Patients undergo allogeneic HCT as in Arm I.
  Patients receive tacrolimus IV or PO on days -1 to 98 (related donor) or 180 (unrelated donor) and mycophenolate mofetil IV over 2 hours or PO every 8 hours on days 1-30 (related donor) or 45 (unrelated donor).
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo allogeneic HCT
  Busulfan: Given IV
  Fludarabine Phosphate: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Mycophenolate Mofetil: Given IV or PO
  Pharmacological Study: Correlative studies
  Tacrolimus: Given IV or PO
- ARM III (Non-Randomized): Patients who were not randomized and did not proceed to transplant because they did not meet all the protocol requirement for randomization
Period: Overall Study
Arm/Group | Arm I (Busulfan, Cyclophosphamide, Melphalan) | Arm II (Busulfan, Fludarabine Phosphate) | ARM III (Non-Randomized)
Started | 6 | 9 | 15
Completed | 5 | 2 | 0
Not Completed | 1 | 7 | 15
Not completed — Death | 0 | 1 | 0
Not completed — Physician Decision | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Progressive Disease | 0 | 5 | 0
Not completed — Ineligible | 0 | 0 | 3
Not completed — No Transplant Planned | 0 | 0 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Busulfan, Cyclophosphamide, Melphalan) | Arm II (Busulfan, Fludarabine Phosphate) | ARM III (Non-Randomized) | Total
Number analyzed (Participants) | 6 | 9 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 9 | 15 | 30
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 0.50 (0.84) | 2.33 (3.71) | 1.27 (1.75) | 1.00 (2.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5 | 10
  Male | 3 | 7 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2 | 4
  Not Hispanic or Latino | 6 | 7 | 13 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 2 | 1 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 3 | 8 | 10 | 21
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 8 | 9 | 23
  Canada | 0 | 0 | 3 | 3
  Australia | 0 | 0 | 1 | 1
  Kuwait | 0 | 1 | 0 | 1
  New Zealand | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Probability of Event-free Survival (EFS)
Description: Probability of Event-free Survival (EFS) for Patients after 18 months. An event is either treatment related mortality (TRM), primary or secondary graft failure, or relapse/non-response (as defined in protocol section 10). Time to event is time from transplant with patients who die between the start of the conditioning regimen and transplant given a time to event of zero.
Time Frame: From transplant up to 18 months
Population: All eligible randomized patients
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Arm I (Busulfan, Cyclophosphamide, Melphalan) | Arm II (Busulfan, Fludarabine Phosphate)
Number analyzed (Participants) | 6 | 9
percent probability | 83 [27 to 97] | 22 [3 to 51]

2. Primary Outcome: Number of Participants Who Experience Treatment-Related Mortality (TRM) by Day 100
Description: The number of patients who experience TRM on day 100. Treatment-Related Mortality (TRM) an event defined as a death prior to relapse or non-response. Time to TRM is defined as time from transplants to TRM. Patients who die between the start of the conditioning regimen and transplant will be considered a TRM with time to TRM of zero.
Time Frame: From transplant up to 100 days
Population: All eligible randomized patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Busulfan, Cyclophosphamide, Melphalan) | Arm II (Busulfan, Fludarabine Phosphate)
Number analyzed (Participants) | 6 | 9
Participants | 0 | 1

3. Secondary Outcome: Percentage of Participants Who Experience Primary Graft Failure Event Between Arms
Description: Primary Graft failure is defined as the failure to achieve an ANC >= 500/uL after 42 days, determined by 3 consecutive measurements on different days; OR < 5% donor cells in blood or bone marrow by day +42 (as demonstrated by a chimerism assay), without evidence of Juvenile Myelomonocytic Leukemia (JMML).
Time Frame: Day 0 - day 540 (18 months) following completion of stem cell transplant
Population: All Eligible randomized patients
Measure: Number; unit: percentage of patients
Arm/Group | Arm I (Busulfan, Cyclophosphamide, Melphalan) | Arm II (Busulfan, Fludarabine Phosphate)
Number analyzed (Participants) | 6 | 9
percentage of patients | 0 | 0

4. Secondary Outcome: Percent Probability of 18 Months-relapse Event Between Arms
Description: Probability of patients relapsing at 18 months. A relapse event is defined in protocol section 10.2.3. Time to relapse/non-response is defined as time from transplant to when all criteria of section 10.2.3 are met.
Time Frame: From transplant up to 18 months
Population: All eligible randomized patients
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Arm I (Busulfan, Cyclophosphamide, Melphalan) | Arm II (Busulfan, Fludarabine Phosphate)
Number analyzed (Participants) | 6 | 9
percent probability | 17 [0.4 to 55] | 55 [16 to 83]

ADVERSE EVENTS:
Time Frame: Up to 1 year after completion of transplant.
Description: Adverse event reporting is collected routinely using case report forms. SAE field contains NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted via expedited reporting (NCI AdEERs / CAeRs). The AE field contains grade 3 and higher CTCAEs reported on study excluding those that were reported as SAEs. Ineligible patients are excluded from reporting of adverse events.
  3 patients from ARM III (Non-Randomized) were excluded due to ineligibility.
Groups:
- ARM III (Non-Randomized): Patients who have not met all protocol requirements to proceed to HCT
Arm/Group | Arm I (Busulfan, Cyclophosphamide, Melphalan) | Arm II (Busulfan, Fludarabine Phosphate) | ARM III (Non-Randomized)
All-Cause Mortality (participants affected / at risk) | 1/6 | 5/9 | 1/12
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/9 | 0/12
Other Adverse Events (participants affected / at risk) | 5/6 | 7/9 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Busulfan, Cyclophosphamide, Melphalan) (N=6) | Arm II (Busulfan, Fludarabine Phosphate) (N=9) | ARM III (Non-Randomized) (N=12)
Multi-organ failure (General disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Busulfan, Cyclophosphamide, Melphalan) (N=6) | Arm II (Busulfan, Fludarabine Phosphate) (N=9) | ARM III (Non-Randomized) (N=12)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (6) | 3 (3) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (4) | 1 (2) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Edema face (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (5) | 3 (3) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (3) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 3 (8) | 1 (1) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (2) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Weight gain (Investigations) | 3 (4) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain sponsor approval

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-05): https://cdn.clinicaltrials.gov/large-docs/93/NCT01824693/Prot_SAP_000.pdf